CLINICAL TRIAL: NCT04409834
Title: A Multicenter, Randomized-Controlled Trial to Evaluate the Efficacy and Safety of Antithrombotic Therapy for Prevention of Arterial and Venous Thrombotic Complications in Critically-Ill COVID-19 Patients
Brief Title: Prevention of Arteriovenous Thrombotic Events in Critically-Ill COVID-19 Patients Trial
Acronym: COVID-PACT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The TIMI Study Group (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CCCTN/TIMI COVID-PACT
Record Dates: First submitted 2020-05-28; First posted 2020-06-01 (Actual); Results first posted 2024-01-19 (Actual); Last update posted 2024-01-19 (Actual); Status verified 2023-12

CONDITIONS: COVID-19; Venous Thromboembolism; Arterial Thrombosis
MeSH Terms: conditions — COVID-19; Venous Thromboembolism | interventions — Enoxaparin; Clopidogrel

STUDY DESIGN:
Intervention Model Description: Randomized-controlled trial - 1) full-dose anticoagulation (FDAC) versus standard-dose prophylactic anticoagulation (SDPAC) (pooled across antiplatelet regimens) and in a subset of patients 2) antiplatelet (AP) versus no AP therapy (pooled across anticoagulant regimens)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Full-dose anticoagulation (FDAC) (Experimental): * Unfractionated heparin (UFH) administered intravenously with a nomogram targeting an activated partial thromboplastin time (aPTT) of 1.5-2.5 times the control as per institutional therapeutic target for treatment of venous thrombotic events (VTE)
  * Enoxaparin 1 mg/kg administered subcutaneously (SC) every 12 hours
  * With or without anti-platelet therapy: Clopidogrel 300 mg administered once orally on the day of randomization, followed by 75 mg administered once daily on subsequent days
  Interventions: Drug: Unfractionated Heparin IV; Drug: Enoxaparin 1 mg/kg; Drug: Clopidogrel
- Standard-dose prophylactic anticoagulation (SDPAC) (Active Comparator): * Enoxaparin 40 mg administered subcutaneously (SC) once daily (reduce to 30 mg if creatinine clearance CrCl <30 ml/min)
  * Heparin 5,000 units administered subcutaneous three times daily
  * With or without anti-platelet therapy: Clopidogrel 300 mg administered once orally on the day of randomization, followed by 75 mg administered once daily on subsequent days
  Interventions: Drug: Clopidogrel; Drug: Unfractionated heparin SC; Drug: Enoxaparin 40 mg SC

INTERVENTIONS:
Drug: Unfractionated Heparin IV — Unfractionated heparin (UFH) administered intravenously with a nomogram targeting an aPTT of 1.5-2.5 times the control as per institutional therapeutic target for treatment of VTE
  Arms: Full-dose anticoagulation (FDAC)
Drug: Enoxaparin 1 mg/kg — Enoxaparin 1 mg/kg administered subcutaneously (SC) every 12 hours
  Other Names: Lovenox
  Arms: Full-dose anticoagulation (FDAC)
Drug: Clopidogrel — Clopidogrel 300 mg administered once orally on the day of randomization, followed by 75 mg administered once daily orally on subsequent days
  Other Names: Plavix
Drug: Unfractionated heparin SC — Heparin 5,000 units administered subcutaneous three times daily
  Arms: Standard-dose prophylactic anticoagulation (SDPAC)
Drug: Enoxaparin 40 mg SC — Enoxaparin 40 mg administered subcutaneously (SC) once daily (reduce to 30 mg if CrCl<30 ml/min)
  Other Names: Lovenox
  Arms: Standard-dose prophylactic anticoagulation (SDPAC)

SUMMARY:
The researchers wanted to learn how to help sick patients who are in the hospital because of COVID-19. They are trying to find out the best way that is safe to stop blood clots that could be dangerous from forming in patients with COVID-19. This research study happened at 34 hospitals.

All patients in the study took medicines that help prevent blood clots. These medicines are called blood thinners or anticoagulants. Patients got different amounts of blood thinners to see what works better and is safer. Researchers randomly chose some patients to get more and some to get less.

The researchers also wanted to know if another medicine called clopidogrel can safely help stop blood clots from forming. This kind of medicine helps keep parts of the blood, called platelets, from sticking together. In some patients who did not have other reasons to take a platelet-blocker the researchers randomly chose the patient to take clopidogrel or not. This type of medicine is also called an antiplatelet.

DETAILED DESCRIPTION:
This is a multicenter, open-label, randomized-controlled trial in critically-ill patients with novel coronavirus disease 2019 (COVID-19) evaluating the efficacy and safety of full-dose vs. standard prophylactic dose anticoagulation and of antiplatelet vs. no antiplatelet therapy (in a nested second randomization) for prevention of venous and arterial thrombotic events. In a subcohort without an ongoing indication for antiplatelet therapy at screening, the second randomization is performed to either antiplatelet or no antiplatelet therapy

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years (male or female)
2. Acute infection with severe acute respiratory syndrome coronavirus 2 (SARS-CoV2)
3. Currently admitted to an intensive care unit (ICU)

Key Exclusion Criteria:

1. Ongoing (>48 hours) or planned full-dose (therapeutic) anticoagulation for any indication
2. Ongoing or planned treatment with dual antiplatelet therapy
3. Contraindication to antithrombotic therapy or high risk of bleeding due to conditions including, but not limited to, any of the following:

   1. History of intracranial hemorrhage, known central nervous system (CNS) tumor or CNS vascular abnormality
   2. Active or recent major bleeding within the past 30 days with untreated source
   3. Platelet count <70,000 or known functional platelet disorder
   4. Fibrinogen <200 mg/dL
   5. International normalized ratio (INR) >1.9
4. History of heparin-induced thrombocytopenia
5. Ischemic stroke within the past 2 weeks

Patients who meet the following criterion are excluded from the second randomization (antiplatelet therapy vs. no antiplatelet therapy):

1. Ongoing or planned antiplatelet therapy, including aspirin monotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 390 (Actual)
Dates: Start 2020-08-05 (Actual); Primary Completion 2022-03-10 (Actual); Study Completion 2022-03-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marc S Sabatine, MD, MPH, Study Chair — The TIMI Study Group; David A Morrow, MD, MPH, Principal Investigator — The TIMI Study Group
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Bohula EA, Berg DD, Lopes MS, Connors JM, Babar I, Barnett CF, Chaudhry SP, Chopra A, Ginete W, Ieong MH, Katz JN, Kim EY, Kuder JF, Mazza E, McLean D, Mosier JM, Moskowitz A, Murphy SA, O'Donoghue ML, Park JG, Prasad R, Ruff CT, Shahrour MN, Sinha SS, Wiviott SD, Van Diepen S, Zainea M, Baird-Zars V, Sabatine MS, Morrow DA; COVID-PACT Investigators. Anticoagulation and Antiplatelet Therapy for Prevention of Venous and Arterial Thrombotic Events in Critically Ill Patients With COVID-19: COVID-PACT. Circulation. 2022 Nov;146(18):1344-1356. doi: 10.1161/CIRCULATIONAHA.122.061533. Epub 2022 Aug 29. PMID 36036760
- [Derived] Fischer AL, Messer S, Riera R, Martimbianco ALC, Stegemann M, Estcourt LJ, Weibel S, Monsef I, Andreas M, Pacheco RL, Skoetz N. Antiplatelet agents for the treatment of adults with COVID-19. Cochrane Database Syst Rev. 2023 Jul 25;7(7):CD015078. doi: 10.1002/14651858.CD015078. PMID 37489818
- [Derived] Lee CK, Merriam LT, Pearson JC, Lipnick MS, McKleroy W, Kim EY. Treating COVID-19: Evolving approaches to evidence in a pandemic. Cell Rep Med. 2022 Feb 9;3(3):100533. doi: 10.1016/j.xcrm.2022.100533. eCollection 2022 Mar 15. PMID 35474746
- [Derived] Flumignan RL, Civile VT, Tinoco JDS, Pascoal PI, Areias LL, Matar CF, Tendal B, Trevisani VF, Atallah AN, Nakano LC. Anticoagulants for people hospitalised with COVID-19. Cochrane Database Syst Rev. 2022 Mar 4;3(3):CD013739. doi: 10.1002/14651858.CD013739.pub2. PMID 35244208

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Patients were randomized in a 1:1 allocation ratio to receive either full-dose anticoagulation (FDAC) or standard-dose prophylactic anticoagulation (SDPAC). In a subset of patients without an ongoing indication for antiplatelet (AP) therapy at baseline, a second randomization was performed in a 1:1 allocation ratio to either AP or no AP therapy. Analyses of anticoagulation were pooled across AP regimens, and AP therapy vs. no AP therapy were pooled across anticoagulant regimens.
Groups:
- Full-dose Anticoagulation (FDAC): * Unfractionated heparin (UFH) administered intravenously with a nomogram targeting an aPTT of 1.5-2.5 times the control as per institutional therapeutic target for treatment of venous thrombotic event (VTE)
  * Enoxaparin 1 mg/kg administered subcutaneously (SC) every 12 hours
  * With or without anti-platelet therapy: Clopidogrel 300 mg administered once orally on the day of randomization, followed by 75 mg administered once daily on subsequent days
- Standard-dose Prophylactic Anticoagulation (SDPAC): * Enoxaparin 40 mg administered subcutaneously (SC) once daily (reduce to 30 mg if creatinine clearance CrCl<30 ml/min)
  * Heparin 5,000 units administered subcutaneous three times daily
  * With or without anti-platelet therapy: Clopidogrel 300 mg administered once orally on the day of randomization, followed by 75 mg administered once daily on subsequent days
Period: Overall Study
Arm/Group | Full-dose Anticoagulation (FDAC) | Standard-dose Prophylactic Anticoagulation (SDPAC)
Started | 197 | 193
Randomized to Anti-platelet Therapy | 74 | 78
Randomized to no Antiplatelet Therapy | 73 | 67
Completed | 142 | 131
Not Completed | 55 | 62
Not completed — Death | 55 | 62

BASELINE CHARACTERISTICS:
Groups:
- Full-dose Anticoagulation (FDAC): * Unfractionated heparin (UFH) administered intravenously with a nomogram targeting an aPTT of 1.5-2.5 times the control as per institutional therapeutic target for treatment of VTE
  * Enoxaparin 1 mg/kg administered subcutaneously(SC) every 12 hours
  * With or without anti-platelet therapy: Clopidogrel 300 mg administered once orally on the day of randomization, followed by 75 mg administered once daily on subsequent days
- Standard-dose Prophylactic Anticoagulation (SDPAC): * Enoxaparin 40 mg administered subcutaneously (SC) once daily (reduce to 30 mg if CrCl<30 ml/min)
  * Heparin 5,000 units administered subcutaneous three times daily
  * With or without anti-platelet therapy: Clopidogrel 300 mg administered once orally on the day of randomization, followed by 75 mg administered once daily on subsequent days
- Total: Total of all reporting groups
Arm/Group | Full-dose Anticoagulation (FDAC) | Standard-dose Prophylactic Anticoagulation (SDPAC) | Total
Number analyzed (Participants) | 197 | 193 | 390
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 59 [51 to 70] | 62 [51 to 68] | 61 [51 to 69]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 75 | 84 | 159
  Male | 122 | 109 | 231
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 135 | 140 | 275
  Non-white | 62 | 53 | 115

OUTCOME MEASURES:

1. Primary Outcome: Venous or Arterial Thrombotic Events: Full-dose Anticoagulation Versus Standard-dose Prophylactic Anticoagulation
Description: The efficacy of these interventions was analyzed using an unmatched win ratio.
  * The number of wins was found by comparing every patient in the FDAC (Full-dose anticoagulation) arm to every patient in the SDPAC (Standard dose prophylactic anticoagulation) arm to determine a 'win' and totaling up the number of wins in each arm.
  * A 'win' is a point in the favor of the arm it is given to. For each comparison of one patient in full dose arm compared to one patient in the standard dose arm, a 'win' is given to arm with the patient who had a component of the composite endpoint either lower in the hierarchy than the paired patient, or if the patient did not have any component of the composite while the paired patient did experience a component event of the composite.
  * Hierarchical composite: Death due to venous or arterial thrombosis, pulmonary embolism, clinically evident DVT, type 1 MI, ischemic stroke, systemic embolism or acute limb ischemia, or clinically silent DVT.
Time Frame: 28 days or until hospital discharge, whichever earlier
Population: The on-treatment analysis population, consisting of all randomly assigned patients who received at least 1 dose of the randomly allocated study strategy. As is pre-specified in the Study Protocol, comparisons between FDAC and SDPAC are reported irrespective of whether participants received anti-platelet therapy.
Measure: Number; unit: Number of wins
Groups:
- Full-dose Anticoagulation: * Unfractionated heparin (UFH) administered intravenously with a nomogram targeting an aPTT of 1.5-2.5 times the control as per institutional therapeutic target for treatment of VTE
  * Enoxaparin 1 mg/kg administered subcutaneously (SC) every 12 hours
- Prophylactic Anticoagulation: * Enoxaparin 40 mg administered SC once daily (reduce to 30 mg if CrCl<30 ml/min)*
  * Heparin 5,000 units administered SC three times daily
Arm/Group | Full-dose Anticoagulation | Prophylactic Anticoagulation
Number analyzed (Participants) | 191 | 191
Number of wins | 4,486 | 2,351
Statistical Analysis 1: Comparison: Full-dose Anticoagulation vs Prophylactic Anticoagulation; FDAC = Full Dose Anticoagulation; SDPAC = Standard Dose Prophylactic Anticoagulation; Test type: Superiority — Stratified Win-Ratio Analysis, 2-sided * The estimated win ratio is calculated by taking the total number of wins in the FDAC arm divided by the total number of wins in the SDPAC arm. A win ratio greater than 1 was in favor of the FDAC arm. * The win ratio methodology is explained in the following reference Pocock et al. Eur Heart J 2012;33:176-82 (doi:10.1093/eurheartj/ehr352); p = 0.028, Stratified Win-Ratio Analysis, 2-sided; Win Ratio = 1.95, 95% CI 2-sided [1.08 to 3.55]

2. Secondary Outcome: Clinically Evident Venous or Arterial Thrombotic Events: Full-dose Anticoagulation Versus Standard-dose Prophylactic Anticoagulation
Description: The efficacy of these interventions was analyzed using an unmatched win ratio.
  * The number of wins was found by comparing every patient in the FDAC (Full-dose anticoagulation) arm to every patient in the SDPAC (Standard dose prophylactic anticoagulation) arm to determine a 'win' and totaling up the number of wins in each arm.
  * A 'win' is a point in the favor of the arm it is given to. For each comparison of one patient in full dose arm compared to one patient in the standard dose arm, a 'win' is given to arm with the patient who had a component of the composite endpoint either lower in the hierarchy than the paired patient, or if the patient did not have any component of the composite while the paired patient did experience a component event of the composite.
  * Hierarchical composite: Death due to venous or arterial thrombosis, pulmonary embolism, clinically evident DVT, type 1 MI, ischemic stroke, systemic embolism or acute limb ischemia.
Time Frame: 28 days or until hospital discharge, whichever earlier
Population: The on-treatment analysis population, consisting of all randomly assigned patients who received at least 1 dose of the randomly allocated study strategy. The on-treatment analysis population, consisting of all randomly assigned patients who received at least 1 dose of the randomly allocated study strategy. As is pre-specified in the Study Protocol, comparisons between FDAC and SDPAC are reported irrespective of whether participants received anti-platelet therapy.
Measure: Number; unit: Number of wins
Groups:
- Prophylactic Anticoagulation: * Enoxaparin 40 mg administered SC once daily (reduce to 30 mg if CrCl<30 ml/min)
  * Heparin 5,000 units administered SC three times daily
Arm/Group | Full-dose Anticoagulation | Prophylactic Anticoagulation
Number analyzed (Participants) | 191 | 191
Number of wins | 3,649 | 2,021
Statistical Analysis 1: Comparison: Full-dose Anticoagulation vs Prophylactic Anticoagulation; FDAC = Full Dose Anticoagulation; SDPAC = Standard Dose Prophylactic Anticoagulation; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.087, Stratified Win-Ratio Analysis, 2-sided; Win Ratio = 1.79, 95% CI 2-sided [0.92 to 3.47]

3. Primary Outcome: Venous or Arterial Thrombotic Events: Anti-platelet Therapy Versus No Anti-platelet Therapy
Description: The efficacy of these interventions was analyzed using an unmatched win ratio.
  * The number of wins was found by comparing every patient in the Anti-platelet group to every patient in the No Anti-platelet group arm to determine a 'win' and totaling up the number of wins in each arm.
  * A 'win' is a point in the favor of the arm it is given to. For each comparison of one patient in full dose arm compared to one patient in the standard dose arm, a 'win' is given to arm with the patient who had a component of the composite endpoint either lower in the hierarchy than the paired patient, or if the patient did not have any component of the composite while the paired patient did experience a component event of the composite.
  * Hierarchical composite: Death due to venous or arterial thrombosis, pulmonary embolism, clinically evident DVT, type 1 MI, ischemic stroke, systemic embolism or acute limb ischemia, or clinically silent DVT.
Time Frame: 28 days or until hospital discharge, whichever earlier
Population: The on-treatment analysis population, consisting of all randomly assigned patients who received at least 1 dose of the randomly allocated study strategy. As is pre-specified in the Study Protocol, comparisons between anti-platelet therapy and no anti-platelet therapy are reported irrespective of which anticoagulation intervention participants received.
Measure: Number; unit: Number of wins
Groups:
- Anti-platelet Therapy: Clopidogrel 300 mg administered once orally on the day of randomization, followed by 75 mg administered once daily on subsequent days.
  Received either FDAC( Unfractionated heparin (UFH) administered intravenously with a nomogram targeting an aPTT of 1.5-2.5 times the control as per institutional therapeutic target for treatment of VTE; or Enoxaparin 1 mg/kg administered subcutaneously (SC) every 12 hours) or SDPAC (Enoxaparin 40 mg administered SC once daily (reduce to 30 mg if CrCl<30 ml/min)*; or Heparin 5,000 units administered SC three times daily).
- No Anti-platelet Therapy: Participants did not receive anti-platelet therapy.
  Received either FDAC( Unfractionated heparin (UFH) administered intravenously with a nomogram targeting an aPTT of 1.5-2.5 times the control as per institutional therapeutic target for treatment of VTE; or Enoxaparin 1 mg/kg administered subcutaneously (SC) every 12 hours) or SDPAC (Enoxaparin 40 mg administered SC once daily (reduce to 30 mg if CrCl<30 ml/min)*; or Heparin 5,000 units administered SC three times daily).
Arm/Group | Anti-platelet Therapy | No Anti-platelet Therapy
Number analyzed (Participants) | 150 | 140
Number of wins | 2052 | 1994
Statistical Analysis 1: Comparison: Anti-platelet Therapy vs No Anti-platelet Therapy; Test type: Superiority — Stratified Win-Ratio Analysis, 2-sided * The estimated win ratio is calculated by taking the total number of wins in the Anti-platelet arm divided by the total number of wins in the No Anti-platelet arm. A win ratio greater than 1 was in favor of the Anti-platelet arm. * The win ratio methodology is explained in the following reference Pocock et al. Eur Heart J 2012;33:176-82 (doi:10.1093/eurheartj/ehr352); p = 0.90, Stratified Win-Ratio Analysis, 2-sided; Win Ratio = 1.04, 95% CI 2-sided [0.54 to 2.01]

4. Secondary Outcome: Clinically Evident Venous or Arterial Thrombotic Events: Anti-platelet Therapy Versus No Anti-platelet Therapy
Description: The efficacy of these interventions was analyzed using an unmatched win ratio.
  * The number of wins was found by comparing every patient in the Anti-platelet group to every patient in the No Anti-platelet group arm to determine a 'win' and totaling up the number of wins in each arm.
  * A 'win' is a point in the favor of the arm it is given to. For each comparison of one patient in full dose arm compared to one patient in the standard dose arm, a 'win' is given to arm with the patient who had a component of the composite endpoint either lower in the hierarchy than the paired patient, or if the patient did not have any component of the composite while the paired patient did experience a component event of the composite.
  * Hierarchical composite: Death due to venous or arterial thrombosis, pulmonary embolism, clinically evident DVT, type 1 MI, ischemic stroke, systemic embolism or acute limb ischemia.
Time Frame: 28 days or until hospital discharge, whichever earlier
Population: as for outcome 3
Measure: Number; unit: Number of wins
Arm/Group | Anti-platelet Therapy | No Anti-platelet Therapy
Number analyzed (Participants) | 150 | 140
Number of wins | 1452 | 1900
Statistical Analysis 1: Comparison: Anti-platelet Therapy vs No Anti-platelet Therapy; Test type: Superiority — [test comment as in outcome 3, analysis 1]; p = 0.53, Stratified Win-Ratio Analysis, 2-sided; Win Ratio = 0.79, 95% CI 2-sided [0.38 to 1.65]

ADVERSE EVENTS:
Time Frame: 28 days or until hospital discharge, whichever earlier
Description: Investigators are required to report: (1) Serious Adverse Events Related to Study Drug, (2) Unexpected Problems, and (3) Adverse Events Leading to Drug Discontinuation.
Groups:
- Antiplatelet Therapy: Clopidogrel 300 mg administered once orally on the day of randomization, followed by 75 mg administered once daily on subsequent days.
- No Anti-platelet Therapy: Participants did not receive anti-platelet therapy.
Arm/Group | Full-dose Anticoagulation (FDAC) | Standard-dose Prophylactic Anticoagulation (SDPAC) | Antiplatelet Therapy | No Anti-platelet Therapy
All-Cause Mortality (participants affected / at risk) | 55/197 | 62/193 | 41/152 | 34/140
Serious Adverse Events (participants affected / at risk) | 16/197 | 3/193 | 6/152 | 0/140
Other Adverse Events (participants affected / at risk) | 37/197 | 22/193 | 25/152 | 0/140
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Full-dose Anticoagulation (FDAC) (N=197) | Standard-dose Prophylactic Anticoagulation (SDPAC) (N=193) | Antiplatelet Therapy (N=152) | No Anti-platelet Therapy (N=140)
Acute Enteritis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Acute Renal Failure (Renal and urinary disorders) | 1 | 0 | 1 | 0
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0
Compartment Syndrome Left Arm (General disorders) | 1 | 0 | 1 | 0
Deep Venous Thrombosis (Vascular disorders) | 0 | 1 | 0 | 0
Drug Induced Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Gastrointestinal bleed (General disorders) | 0 | 1 | 0 | 0
Gross Hematuria (General disorders) | 1 | 0 | 1 | 0
Hematemesis (General disorders) | 1 | 0 | 0 | 0
Intracranial Hemmorrhage (General disorders) | 1 | 0 | 0 | 0
Lower Respiratory Tract Bleed (General disorders) | 1 | 0 | 1 | 0
Pulmonary bleeding from left upper lobe (General disorders) | 1 | 0 | 0 | 0
Rectus Sheath Hematoma (General disorders) | 1 | 0 | 0 | 0
Retroperitoneal Bleed (General disorders) | 1 | 1 | 1 | 0
Retroperitoneal hematoma (General disorders) | 3 | 0 | 1 | 0
Right Rectus Intramuscular Hematoma (General disorders) | 1 | 0 | 1 | 0
Right upper extremity soft tissue hematoma (General disorders) | 1 | 0 | 0 | 0
Right wrist intramural hematoma (General disorders) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Full-dose Anticoagulation (FDAC) (N=197) | Standard-dose Prophylactic Anticoagulation (SDPAC) (N=193) | Antiplatelet Therapy (N=152) | No Anti-platelet Therapy (N=140)
Bleeding (General disorders) | 35 | 3 | 23 | 0
Venous thromboembolism (Vascular disorders) | 2 | 9 | 2 | 0
D-dimer elevation (Blood and lymphatic system disorders) | 0 | 10 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-10-28): https://cdn.clinicaltrials.gov/large-docs/34/NCT04409834/Prot_SAP_000.pdf